CLINICAL TRIAL: NCT00774982
Title: Pilot, Randomized, Open-Label, Two-Way Crossover Comparative Bioavailability Study of 40 mg Delayed Release Oral 6Mercaptopurine Versus 100 mg Purinethol in Patients With Crohns Disease
Brief Title: Pilot Comparative Bioavailability Study of 6Mercaptopurine (Delayed Release vs. Purinethol) in Crohns Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva GTC (Industry)
Responsible Party: Prof. Yaron Ilan, Hadasssah Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: C1/13/6MP-02
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Crohns Disease
Keywords: Crohns Disease; Pharmacokinetics; Local Targeted Delivery to the Ileum; Delayed Release; Immunology Measurements; Pharmacokinetics in Crohns Disease Patients
MeSH Terms: conditions — Crohn Disease | interventions — Mercaptopurine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 6MP Test Formulation (Experimental): 1 x 40 mg Oral Tablet, 6 MP Delayed Release Test Formulation, for targeted ileal delivery
  Interventions: Drug: Delayed Release 6 mercaptopurine
- 2. 6MP Reference Formulation (Active Comparator): 2 x 50 mg oral tablet, PURINETHOL
  Interventions: Drug: 6 Mercaptopurine

INTERVENTIONS:
Drug: Delayed Release 6 mercaptopurine — oral tablet, 1 x 40 mg Delayed Release 6MP tablet, single-dose
  Other Names: Administration 1 (A): 1 x 40 mg Delayed Release 6MP TEST
  Arms: 1 6MP Test Formulation
Drug: 6 Mercaptopurine — Oral Tablet, 2 x 50 mg 6MP Reference, single-dose
  Other Names: Administration 2 (B): 2 x 50 mg Purinethol REFERENCE
  Arms: 2. 6MP Reference Formulation

SUMMARY:
The study is being conducted to evaluate the pharmacokinetic parameters (Cmax, Tmax and AUC) of the new delayed release, lowered dose, 40 mg 6MP test formulation as compared to standard 6MP (100 mg Purinethol) in 12 patients with Crohn's Disease.

The study is being undertaken to prove that the new test formulation is indeed delayed-release and targeted to the ileum, and that the levels of 6MP in the blood following local absorption are lower than that seen following standard Purinethol dosing. This should result in lower, safer mercaptopurine dosing, allowing for uninterrupted treatment with fewer side effects.

DETAILED DESCRIPTION:
A new delayed release, faster-disintegrating, lower dose oral formulation of 6 mercaptopurine for targeted delivery to the ileum (the most commonly effected area of Crohns Disease (CD) bowel involvement), was developed and shown to be effective in the three efficacy parameters evaluated in a small group of Crohns Disease patients. Twelve weeks of daily treatment with once-nightly dosing of 40 mg local 6MP resulted in: (1) inducing clinical remission (CDAI scores below 150 as early as weeks 2 and 4), (2) effecting local mucosal healing (as evidenced by lowered CDEIS scores and descriptive conolonoscopy reports) and (3) reducing systemic immunological scores (lowered IFN-gamma Elispot levels).

The current study is being undertaken to confirm, via pharmacokinetic profiles (Cmax, AUC and Tmax), the underlying premises of the above-noted clinical feasibility study. This PK study is being conducted to establish that (1) The delayed release test formulation delivers drug distally to the lower intestine and (2) The delayed release test formulation has the potential for reduced systemic toxicity. The first aspect will be established by comparing the Tmax of the delayed release test formulation vs. oral Purinethol, while the second aspect will be established by comparing the Cmax and AUC of the 40 mg test dose vs. standard 100 mg Purinethol. It is anticipated that the delayed release test formulation will exhibit a later Tmax and reduced Cmax and AUC as compared to reference Purinethol.

Additionally, immunology testing to measure the effect of the new 6MP formulation on immunological FACS analysis will be performed on peripheral blood lymphocytes at 0, 12 and 24 hours post-dosing of each formualtion. Lymphocytes will be tested for surface marker expression (ex: CD3, CD4, CD8, CD25, NKT, etc.), with anticipated results a greater lowering of immune parameters after even 1 dose of 40 mg delayed release test drug, as compared to 100 mg Purinethol.

ELIGIBILITY:
Inclusion Criteria:

* 12 male and non-pregnant females, aged 18-50 years, with Crohns Disease (CDAI up to 200), non-smoking.

Crohns Disease diagnosis via colonoscopy with biopsy within the past 12 years No CD medications allowed during study other than 5-ASA and symptomatic relief (anti-diarrheals) Screening lab tests: HGB>= 8.5 g/dl, platelets >= 100,000/mm3, WBC: 3500-12000/mm3, serum albumin above 2.5 g/dl, amylase, lipase and total bilirubin within normal limits; ALT, AST, alkaline phosphatase up to 1.5 x normal limits

Exclusion Criteria:

* No more than 2 bowel movements/24 hour period in week prior to screening No patients on methotrexate, cyclosporine, or other anti-TNF alpha, or anti-neoplastics within 3 months of study start NO fistulizing CD or isolated small bowle CD No symptomatic stenosis or ileal strictures,or x-ray evidnece of fibrosed bowel

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
PK parameters: AUC, Cmax and Tmax | Following single dose of test or reference drug

SECONDARY OUTCOMES:
FACS analysis of peripheral blood lymphocytes following single dose of test vs. reference formulation | Comparison of values from blood collected at 0, 12 and 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel